CLINICAL TRIAL: NCT05911529
Title: Motivational Interviewing for Patients With Acute Psychosis
Acronym: MIA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Psychiatric University Hospital, Zurich (Other)
Responsible Party: Principal Investigator, Rahel Horisberger, Clinical psychologist, PhD, Psychiatric University Hospital, Zurich
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MI for acute psychosis
Record Dates: First submitted 2023-05-02; First posted 2023-06-22 (Actual); Last update posted 2024-07-16 (Actual); Status verified 2024-07

CONDITIONS: Psychosis; Schizophrenia
Keywords: Psychosis; Motivational Interviewing; Psychotherapy for psychosis; Adherence to treatment; Therapeutic alliance; Acute phase
MeSH Terms: conditions — Psychotic Disorders; Schizophrenia; Treatment Adherence and Compliance | interventions — Motivational Interviewing

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Motivational Interviewing Group (Experimental): Patients will receive four sessions of Motivational Interviewing within two weeks.
  Interventions: Behavioral: Motivational Interviewing
- Control Group (Active Comparator): Patients in the control group receive four sessions of supportive conversations within two weeks.
  Interventions: Behavioral: Supportive conversations

INTERVENTIONS:
Behavioral: Motivational Interviewing — In our study intervention, patients should receive four session of motivational interviewing (MI). Throughout the MI sessions, interviewers use common MI techniques including open-ended questions, affirmations, reflections, summaries, asking permission, expressing empathy, supporting self-efficacy, etc. Interviewers are clinical psychologists who received MI training immediately prior to the study.
  Arms: Motivational Interviewing Group
Behavioral: Supportive conversations — In the control intervention patients should also be given four sessions, in which no MI techniques take place. They will be carried out in the sense of supportive conversations (i. e. conver-sations that do not follow a specific psychotherapy concept).
  Since we want to check whether the patients really benefit from the specific intervention and not from getting more speaking time, the patient in the control group will also be given four conver-sations. It is known that supportive conversations can have a certain effect on the well-being and recovery process of patients, as the therapeutic relationship, i.e. appreciation, attention and/or attention, is an important efficacy factor (e. g. Grawe, 1995).
  Arms: Control Group

SUMMARY:
Psychotic disorders are associated with high levels of distress, limitations in quality of life, and a high risk of chronification for those affected. The treatment guidelines recommend combining the pharmacological treatment with psychotherapeutic methods, starting already in the acute phase. At the same time, there is little research evidence on which mechanisms of psychotherapy are most effective and best feasible for the acute setting. Therefore, the aim is to run a pilot study to test specific psychotherapeutic interventions for patients with psychosis on acute psychiatric wards.

The method of "Motivational Interviewing" is a well-known and established interviewing technique, which originally comes from the treatment of addictive disorders. In this study, it is used to strengthen the therapeutic alliance between patient and practitioner already in the acute phase of the disease, to increase adherence, and thus to achieve the overall goal of better integrating patients with pronounced positive symptoms into treatment. This appears to be extremely important, as non-adherence represents one of the greatest risks for chronification of the disease. The intervention will subsequently be evaluated in comparison to "treatment as usual".

DETAILED DESCRIPTION:
Psychotic disorders are among the top ten causes of long-term disability and have a high chronicity potential and a high risk of invalidity. One-fifth of all patients with schizophrenia suffer from chronic symptoms and impairments, and the disease is associated with low long-term work performance, a high degree of all mental health care resources and high socioeconomic costs. These findings demonstrate the importance of sufficient treatment for psychotic disorders and, most importantly, point to a need for research so that more effective treatments can be developed in the future.

In the recent decade, various psychotherapeutic programs with cognitive-behavioral background have been developed for patients with psychosis, and their efficacy has been investigated. Meta-analyses have shown superiority of cognitive-behavioral therapy for psychosis over standard treatment, both in combination with antipsychotic medication and without. Many of the psychological approaches have focused primarily on treating the deficits associated with psychosis, as for example cognitive remediation or social skills training. However, these methods are not feasible in the acute setting and there are only a few psychotherapeutic instruments that can be used within a short period of time for inpatient treatment.

The guidelines for the treatment of schizophrenia recommend a combination of antipsychotic medication and psychosis-specific cognitive behavioral therapy. This includes all stages of the illness, also in the acute phase. The Swiss Society for Psychiatry and Psychotherapy (SGPP) has stated in its treatment guidelines for schizophrenia that "our group recommends a structured psychotherapeutic approach even in the acute phase of the disease. The best evidence currently exists for cognitive-behavioral approaches, […]. In any case, the psychotherapeutic procedure must be adapted to the circumstances of the acute phase and there is an urgent need for research on how this can be arranged in the setting of an acute ward.". Despite this explicit recommendation, to our knowledge there have been no studies that have systematically investigated this in the acute setting and results of which could therefore inform future treatment recommendations. As proposed by the SGPP, the aim is to systematically test and evaluate psychotherapeutic interventions in the setting of an acute care unit in an initial pilot trial.

Therapeutic alliance during the acute phase of psychotic illness is one of the most pressing obstacles for successful long term recovery. In order for patients to accept much-needed medication and psychosocial therapy and not drop out prematurely, intrinsic motivation to adhere to therapy is crucial. Motivational Interviewing is a method, that has been developed and evaluated over the last three decades and that shows promising results, not only for patients with addiction but also for other patients who struggle with compliance and ambivalence towards treatment and change of behavior.

It is well known from clinical experience that patients are offered psychotherapy only late during the course of hospitalizations and not when it is highly needed - during the acute phase of their illness. Accordingly, there is a clear gap in the literature as to which interventions are particularly useful in this challenging yet crucial phase of the illness.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent as documented by signature
* Male and female patients from inpatient units of the Psychiatric University Hospital of Zurich
* ICD-10 diagnosis of psychosis (F2.x)
* Fluent in German and able to understand the instructions

Exclusion Criteria:

* Organic schizophrenia-like disorder (ICD: F0.6)
* Drug or alcohol abuse during treatment
* Previous enrolment in the current study
* Enrolment of the investigator, his/her family members, employees and other dependent persons
* During study: Complete stop of taking antipsychotic medications

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2023-03-15 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Change from Baseline in Therapeutic Alliance on the Scale to Assess Therapeutic Relationship | Baseline and week 3 (or after 4 sessions of psychotherapeutic intervention)
  The therapeutic relationship will be evaluated with the german version of the Scale to Assess Therapeutic Relationship (STAR). The patient (STAR-P) and clinician scales (STAR-C) each have 12 items comprising three subscales: positive collaboration and posi-tive clinician input in both versions, non-supportive clinician input in the patient version, and emotional difficulties in the clinician version.
Change from Baseline in Treatment Adherence on the Brief Adherence Rating Scale | Baseline and week 3 (or after 4 sessions of psychotherapeutic intervention)
  The Brief Adherence Rating Scale (BARS) is a brief, pencil-paper, clinician-administered adherence assessment instrument. It consists of 4 items: 3 questions and an overall visual analog rating scale to assess the proportion of doses taken by the patient in the past month (0%-100%).

SECONDARY OUTCOMES:
Change from Baseline in Symptom Severity measured with the Positive and Negative Syndrome Scale | Baseline and week 3 (or after 4 sessions of psychotherapeutic intervention)
  Psychotic symptoms are assessed with the Positive and Negative Syndrome Scale (PANSS). This is a structured interview, which consists of four scales measuring positive and negative syndromes of schizophrenia, their differential, and general severity of illness.
Change from Baseline in Motivation for psychotherapy in the Questionnaire to measure the motivation for psychotherapy | Baseline and week 3 (or after 4 sessions of psychotherapeutic intervention)
  Motivation for psychotherapy will be measured with the german version of the Questionnaire to measure the motivation for psychotherapy, a 4-point Likert-scale with 39 items.
Change from Baseline in Self-Efficacy on the General Self-Efficacy Scale | Baseline and week 3 (or after 4 sessions of psychotherapeutic intervention)
  Self-efficacy is measured with the german version of the General Self-Efficacy Scale (GSE), an instrument that has been proved with a sample of more than 19'000 persons in 25 countries and shows good psychometric properties.

CONTACTS AND LOCATIONS:
Overall Officials: Philipp Homan, Prof., Principal Investigator — University of Zurich
Locations (1):
- Psychiatric University Hospital Zurich, Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] McGuire-Snieckus R, McCabe R, Catty J, Hansson L, Priebe S. A new scale to assess the therapeutic relationship in community mental health care: STAR. Psychol Med. 2007 Jan;37(1):85-95. doi: 10.1017/S0033291706009299. Epub 2006 Nov 9. PMID 17094819
- [Background] Kay SR, Fiszbein A, Opler LA. The positive and negative syndrome scale (PANSS) for schizophrenia. Schizophr Bull. 1987;13(2):261-76. doi: 10.1093/schbul/13.2.261. PMID 3616518
- [Background] Byerly MJ, Nakonezny PA, Rush AJ. The Brief Adherence Rating Scale (BARS) validated against electronic monitoring in assessing the antipsychotic medication adherence of outpatients with schizophrenia and schizoaffective disorder. Schizophr Res. 2008 Mar;100(1-3):60-9. doi: 10.1016/j.schres.2007.12.470. Epub 2008 Feb 5. PMID 18255269
- [Background] Schwarzer, R., & Jerusalem, M. (1995). Generalized self-efficacy scale. In J. Weinman, S. Wright, & M. Johnston, Measures in health psychology: A user's portfolio causal and control beliefs. (pp. 35-37). NFER-NELSON.
- [Background] Schulz, H., Nübling, R., & Rüddel, H. (1995). Entwicklung einer Kurzform eines Fragebogens zur Psychotherapiemotivation. Verhaltenstherapie, 5, 89-95.
- [Background] Aghotor J, Pfueller U, Moritz S, Weisbrod M, Roesch-Ely D. Metacognitive training for patients with schizophrenia (MCT): feasibility and preliminary evidence for its efficacy. J Behav Ther Exp Psychiatry. 2010 Sep;41(3):207-11. doi: 10.1016/j.jbtep.2010.01.004. Epub 2010 Jan 28. PMID 20167306
- [Background] Bark N, Revheim N, Huq F, Khalderov V, Ganz ZW, Medalia A. The impact of cognitive remediation on psychiatric symptoms of schizophrenia. Schizophr Res. 2003 Oct 1;63(3):229-35. doi: 10.1016/s0920-9964(02)00374-2. PMID 12957702
- [Background] Cavelti M, Homan P, Vauth R. The impact of thought disorder on therapeutic alliance and personal recovery in schizophrenia and schizoaffective disorder: An exploratory study. Psychiatry Res. 2016 May 30;239:92-8. doi: 10.1016/j.psychres.2016.02.070. Epub 2016 Mar 2. PMID 27137967
- [Background] Galderisi S, Kaiser S, Bitter I, Nordentoft M, Mucci A, Sabe M, Giordano GM, Nielsen MO, Glenthoj LB, Pezzella P, Falkai P, Dollfus S, Gaebel W. EPA guidance on treatment of negative symptoms in schizophrenia. Eur Psychiatry. 2021 Mar 17;64(1):e21. doi: 10.1192/j.eurpsy.2021.13. PMID 33726883
- [Background] Grawe, K. (1995). Grundriss einer Allgemeinen Psychotherapie. Psychotherapeut, 40, 130-145.
- [Background] Kahn RS, Sommer IE, Murray RM, Meyer-Lindenberg A, Weinberger DR, Cannon TD, O'Donovan M, Correll CU, Kane JM, van Os J, Insel TR. Schizophrenia. Nat Rev Dis Primers. 2015 Nov 12;1:15067. doi: 10.1038/nrdp.2015.67. PMID 27189524
- [Background] Kaiser, S., Berger, G., Conus, P., Kawohl, W., Müller, T. J., Schimmelmann, B. G., Traber, R., Trächsel, N., Vauth, R., & Seifritz, E. (2016). SGPP Behandlungsempfehlungen Schizophrenie. Schweizerische Gesellschaft für Psychiatrie und Psychotherapie.
- [Background] Kennedy JL, Altar CA, Taylor DL, Degtiar I, Hornberger JC. The social and economic burden of treatment-resistant schizophrenia: a systematic literature review. Int Clin Psychopharmacol. 2014 Mar;29(2):63-76. doi: 10.1097/YIC.0b013e32836508e6. PMID 23995856
- [Background] Kuipers E, Yesufu-Udechuku A, Taylor C, Kendall T. Management of psychosis and schizophrenia in adults: summary of updated NICE guidance. BMJ. 2014 Feb 12;348:g1173. doi: 10.1136/bmj.g1173. No abstract available. PMID 24523363
- [Background] Lincoln, T. M., & Pedersen, A. (2019). An Overview of the Evidence for Psychological Interventions for Psychosis: Results From Meta-Analyses. Clinical Psychology in Europe, 1(1), 1-23. https://doi.org/10.32872/cpe.v1i1.31407
- [Background] Mehl, S., & Lincoln, T. (2014). Therapie-Tools Psychose. Beltz.
- [Background] Morrison AP, Hutton P, Wardle M, Spencer H, Barratt S, Brabban A, Callcott P, Christodoulides T, Dudley R, French P, Lumley V, Tai SJ, Turkington D. Cognitive therapy for people with a schizophrenia spectrum diagnosis not taking antipsychotic medication: an exploratory trial. Psychol Med. 2012 May;42(5):1049-56. doi: 10.1017/S0033291711001899. Epub 2011 Sep 14. PMID 21914252
- [Background] Morrison AP, Turkington D, Pyle M, Spencer H, Brabban A, Dunn G, Christodoulides T, Dudley R, Chapman N, Callcott P, Grace T, Lumley V, Drage L, Tully S, Irving K, Cummings A, Byrne R, Davies LM, Hutton P. Cognitive therapy for people with schizophrenia spectrum disorders not taking antipsychotic drugs: a single-blind randomised controlled trial. Lancet. 2014 Apr 19;383(9926):1395-403. doi: 10.1016/S0140-6736(13)62246-1. Epub 2014 Feb 6. PMID 24508320
- [Background] Mueser KT, McGurk SR. Schizophrenia. Lancet. 2004 Jun 19;363(9426):2063-72. doi: 10.1016/S0140-6736(04)16458-1. PMID 15207959
- [Background] Murray, C. J. L., & Lopez, A. D. (1996). The global burden of disease: a comprehensive assessment of mortality and disability from diseases, injuries, and risk factors in 1990 and projected to 2020.
- [Background] National Institute for Health and Clinical Excellence (2010). Schizophrenia: The NICE Guideline on Core Interventions in the Treatment and Management of Schizophrenia in Adults in Primary and Secondary Care. http://www.nice.org.uk/nicemedia/pdf/CG82FullGuideline.pdf
- [Background] Owen MJ, Sawa A, Mortensen PB. Schizophrenia. Lancet. 2016 Jul 2;388(10039):86-97. doi: 10.1016/S0140-6736(15)01121-6. Epub 2016 Jan 15. PMID 26777917
- [Background] Puig O, Penades R, Baeza I, De la Serna E, Sanchez-Gistau V, Bernardo M, Castro-Fornieles J. Cognitive remediation therapy in adolescents with early-onset schizophrenia: a randomized controlled trial. J Am Acad Child Adolesc Psychiatry. 2014 Aug;53(8):859-68. doi: 10.1016/j.jaac.2014.05.012. Epub 2014 Jun 21. PMID 25062593
- [Background] Rabinowitz J, Levine SZ, Garibaldi G, Bugarski-Kirola D, Berardo CG, Kapur S. Negative symptoms have greater impact on functioning than positive symptoms in schizophrenia: analysis of CATIE data. Schizophr Res. 2012 May;137(1-3):147-50. doi: 10.1016/j.schres.2012.01.015. Epub 2012 Feb 6. PMID 22316568

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-02-10): https://cdn.clinicaltrials.gov/large-docs/29/NCT05911529/Prot_SAP_000.pdf